CLINICAL TRIAL: NCT02699411
Title: Dry Needling Effectiveness of Patients on Break Anterior Cruciate Ligament. Single-Blind Randomized Clinical Trial.
Brief Title: Dry Needling Effectiveness of Patients on Break Anterior Cruciate Ligament.
Acronym: ACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European University Spain (Other)
Responsible Party: Principal Investigator, Jorge Velázquez Saornil, Physiotherapist, European University Spain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: European University
Record Dates: First submitted 2016-02-26; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: ligament anterior cruciate , dry needling, physioterapy, propioception, knee arthroplasty, vastus medialis.
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dry needling (Active Comparator): Dry needling on the vastus is performed in patients undergoing ACL fortnight after the intervention and then evaluated. REL dry needling while supplies last twenty insertions before treatment, at midnight, a week and five weeks.
  Interventions: Device: Dry needling
- Stability and propioception (Active Comparator): Proprioception and stability exercises in patients undergoing ACL fortnight after the intervention and then evaluates performed before treatment, at midnight, a week and five weeks.
  Interventions: Other: Stability and propioception

INTERVENTIONS:
Device: Dry needling — dry needling Travell and Simons
  Arms: dry needling
Other: Stability and propioception — Start excursion balance test, WOMAC; ROM, EVA.
  Arms: Stability and propioception

SUMMARY:
We will conduct a randomized clinical trial observing forty patients divided into two groups: one group composed of twenty individuals undergoing surgery for ruptured ACL, which perform dry needling of myofascial trigger (PGM) point of the vastus muscle and then perform techniques proprioception (group a); and twenty patients not be treated with dry needling after ACL surgery, using only proprioceptive exercises to the joint (group B).

DETAILED DESCRIPTION:
It carries out a last fifteen days ECA surgical reconstruction of the anterior cruciate ligament. Twenty individuals in a group to be subjected to a technique of physiotherapy, dry needling were included. (Group A). Another group of twenty patients treated with conservative treatment performed a stability exercises and proprioception (Group B). Forty-six patients will be examined s. None had been previously operated by joint instability and all subjects were previously subjected to a diagnostic study by nuclear magnetic resonance before surgery and the diagnosis was confirmed by additional diagnostic testing. All patients will be evaluated by a physical therapist and Myofascial Trigger Point (PGM) of the vastus muscle will be evaluated.

patients using the following variables are evaluated:

* Pain: Visual Analog Scale (VAS) was used.
* Stiffness and physical function using the WOMAC scale (The Western Ontario and McMaster Universities Arthritis Index.).
* Range of motion of the knee joint: Scale ROM.
* Muscular strength, balance and propiocepción: Star Excursion by Balance Scale Test.

ELIGIBILITY:
Inclusion Criteria:

* over eighteen and anatomically mature surgically break LCA and valued above using MRI and functional tests to confirm the rupture of the ligament.

Exclusion Criteria:

* Patients who did not reach 18 years of age and those over 55,
* postoperative complications
* cause myofascial or neuropathic pain in the lower limb, as lumba-sacral radiculopathy, neuropraxia, neurotmesis, axonotmesis or meralgia paresthetica;
* fibromyalgia.
* hypothyroidism
* iron deficiencies and patients who had a fear of needles (fear of needles).
* Lower limb differences.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Degree range of motion (ROM) | 24 hours
Scores ofThe Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 24 hours
Pain scores visual analog scale (EVA) | 24 hours
Scores of STAR BALANCE TEST | 24

SECONDARY OUTCOMES:
Degree range of motion (ROM) | 1 week
Degree range of motion (ROM) | 5 weeks
Scores ofThe Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 1 week
Scores ofThe Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 5 weeks
Pain scores visual analog scale (EVA) | 1 week
Pain scores visual analog scale (EVA) | 5 weeks
Scores STAR BALANCE TEST | 1week
Scores STAR BALANCE TEST | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Velázquez, Sr, Principal Investigator — European University
Locations (1):
- Jorge Velázquez Saornil, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adachi N, Ochi M, Uchio Y, Iwasa J, Ryoke K, Kuriwaka M. Mechanoreceptors in the anterior cruciate ligament contribute to the joint position sense. Acta Orthop Scand. 2002 Jun;73(3):330-4. doi: 10.1080/000164702320155356. PMID 12143983
- [Background] Ahn JH, Chang MJ, Lee YS, Koh KH, Park YS, Eun SS. Non-operative treatment of ACL rupture with mild instability. Arch Orthop Trauma Surg. 2010 Aug;130(8):1001-6. doi: 10.1007/s00402-010-1077-4. Epub 2010 Mar 25. PMID 20336305
- [Background] Alentorn-Geli E, Myer GD, Silvers HJ, Samitier G, Romero D, Lazaro-Haro C, Cugat R. Prevention of non-contact anterior cruciate ligament injuries in soccer players. Part 1: Mechanisms of injury and underlying risk factors. Knee Surg Sports Traumatol Arthrosc. 2009 Jul;17(7):705-29. doi: 10.1007/s00167-009-0813-1. Epub 2009 May 19. PMID 19452139
- [Background] Domingo A, Mayoral O, Monterde S, Santafe MM. Neuromuscular damage and repair after dry needling in mice. Evid Based Complement Alternat Med. 2013;2013:260806. doi: 10.1155/2013/260806. Epub 2013 Apr 9. PMID 23662122
- [Background] Baltaci G, Harput G, Haksever B, Ulusoy B, Ozer H. Comparison between Nintendo Wii Fit and conventional rehabilitation on functional performance outcomes after hamstring anterior cruciate ligament reconstruction: prospective, randomized, controlled, double-blind clinical trial. Knee Surg Sports Traumatol Arthrosc. 2013 Apr;21(4):880-7. doi: 10.1007/s00167-012-2034-2. Epub 2012 Apr 29. PMID 22543515
- [Background] Sbihi A, Franceschi JP, Christel P, Colombet P, Djian P, Bellier G. [Anterior cruciate ligament reconstruction: biomechanical comparison on cadaver specimens using a single or double hamstring technique]. Rev Chir Orthop Reparatrice Appar Mot. 2004 Nov;90(7):643-50. doi: 10.1016/s0035-1040(04)70725-4. French. PMID 15625515
- [Background] Caraffa A, Cerulli G, Projetti M, Aisa G, Rizzo A. Prevention of anterior cruciate ligament injuries in soccer. A prospective controlled study of proprioceptive training. Knee Surg Sports Traumatol Arthrosc. 1996;4(1):19-21. doi: 10.1007/BF01565992. PMID 8963746
- [Background] Cimino F, Volk BS, Setter D. Anterior cruciate ligament injury: diagnosis, management, and prevention. Am Fam Physician. 2010 Oct 15;82(8):917-22. PMID 20949884
- [Background] Delince P, Ghafil D. Anterior cruciate ligament tears: conservative or surgical treatment? Knee Surg Sports Traumatol Arthrosc. 2013 Jul;21(7):1706-7. doi: 10.1007/s00167-012-2134-z. Epub 2012 Jul 13. No abstract available. PMID 22790441
- [Background] Diekstall P, Rauhut F. [Considerations for the indications for anterior cruciate ligament reconstruction. Results of conservative versus operative treatment]. Unfallchirurg. 1999 Mar;102(3):173-81. doi: 10.1007/s001130050390. German. PMID 10232033
- [Background] Dommerholt J. Dry needling - peripheral and central considerations. J Man Manip Ther. 2011 Nov;19(4):223-7. doi: 10.1179/106698111X13129729552065. PMID 23115475
- [Background] Fithian DC, Paxton EW, Stone ML, Luetzow WF, Csintalan RP, Phelan D, Daniel DM. Prospective trial of a treatment algorithm for the management of the anterior cruciate ligament-injured knee. Am J Sports Med. 2005 Mar;33(3):335-46. doi: 10.1177/0363546504269590. PMID 15716249
- [Background] Fitzgerald GK, Axe MJ, Snyder-Mackler L. The efficacy of perturbation training in nonoperative anterior cruciate ligament rehabilitation programs for physical active individuals. Phys Ther. 2000 Feb;80(2):128-40. PMID 10654060
- [Background] Friederich NF, O'Brien WR. [Gonarthrosis after injury of the anterior cruciate ligament: a multicenter, long-term study]. Z Unfallchir Versicherungsmed. 1993;86(2):81-9. German. PMID 8251257
- [Background] Garvey TA, Marks MR, Wiesel SW. A prospective, randomized, double-blind evaluation of trigger-point injection therapy for low-back pain. Spine (Phila Pa 1976). 1989 Sep;14(9):962-4. doi: 10.1097/00007632-198909000-00008. PMID 2528826
- [Background] Gelb HJ, Glasgow SG, Sapega AA, Torg JS. Magnetic resonance imaging of knee disorders. Clinical value and cost-effectiveness in a sports medicine practice. Am J Sports Med. 1996 Jan-Feb;24(1):99-103. doi: 10.1177/036354659602400118. PMID 8638763
- [Background] Basdekis G, Christel P, Anne F. Validation of the position of the femoral tunnels in anatomic double-bundle ACL reconstruction with 3-D CT scan. Knee Surg Sports Traumatol Arthrosc. 2009 Sep;17(9):1089-94. doi: 10.1007/s00167-009-0829-6. Epub 2009 Jun 13. PMID 19526223
- [Background] Harris JD, Erickson BJ, Bach BR Jr, Abrams GD, Cvetanovich GL, Forsythe B, McCormick FM, Gupta AK, Cole BJ. Return-to-Sport and Performance After Anterior Cruciate Ligament Reconstruction in National Basketball Association Players. Sports Health. 2013 Nov;5(6):562-8. doi: 10.1177/1941738113495788. PMID 24427434
- [Background] Hewett TE, Myer GD, Ford KR, Heidt RS Jr, Colosimo AJ, McLean SG, van den Bogert AJ, Paterno MV, Succop P. Biomechanical measures of neuromuscular control and valgus loading of the knee predict anterior cruciate ligament injury risk in female athletes: a prospective study. Am J Sports Med. 2005 Apr;33(4):492-501. doi: 10.1177/0363546504269591. Epub 2005 Feb 8. PMID 15722287
- [Background] Jinks C, Jordan K, Croft P. Measuring the population impact of knee pain and disability with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Pain. 2002 Nov;100(1-2):55-64. doi: 10.1016/s0304-3959(02)00239-7. PMID 12435459
- [Background] Koga H, Nakamae A, Shima Y, Iwasa J, Myklebust G, Engebretsen L, Bahr R, Krosshaug T. Mechanisms for noncontact anterior cruciate ligament injuries: knee joint kinematics in 10 injury situations from female team handball and basketball. Am J Sports Med. 2010 Nov;38(11):2218-25. doi: 10.1177/0363546510373570. Epub 2010 Jul 1. PMID 20595545
- [Background] Krosshaug T, Nakamae A, Boden BP, Engebretsen L, Smith G, Slauterbeck JR, Hewett TE, Bahr R. Mechanisms of anterior cruciate ligament injury in basketball: video analysis of 39 cases. Am J Sports Med. 2007 Mar;35(3):359-67. doi: 10.1177/0363546506293899. Epub 2006 Nov 7. PMID 17092928
- [Background] Johnson RJ, Beynnon BD. What do we really know about rehabilitation after ACL reconstruction?: commentary on an article by L.M. Kruse, MD, et al.: "rehabilitation after anterior cruciate ligament reconstruction. a systematic review". J Bone Joint Surg Am. 2012 Oct 3;94(19):e148(1-2). doi: 10.2106/JBJS.L.00947. No abstract available. PMID 23032598
- [Background] Lephart SM, Pincivero DM, Giraldo JL, Fu FH. The role of proprioception in the management and rehabilitation of athletic injuries. Am J Sports Med. 1997 Jan-Feb;25(1):130-7. doi: 10.1177/036354659702500126. PMID 9006708
- [Background] Li G, DeFrate LE, Sun H, Gill TJ. In vivo elongation of the anterior cruciate ligament and posterior cruciate ligament during knee flexion. Am J Sports Med. 2004 Sep;32(6):1415-20. doi: 10.1177/0363546503262175. Epub 2004 Jul 20. PMID 15310565
- [Background] Orishimo KF, Liederbach M, Kremenic IJ, Hagins M, Pappas E. Comparison of landing biomechanics between male and female dancers and athletes, part 1: Influence of sex on risk of anterior cruciate ligament injury. Am J Sports Med. 2014 May;42(5):1082-8. doi: 10.1177/0363546514523928. Epub 2014 Mar 3. PMID 24590005
- [Background] Liu-Ambrose T, Taunton JE, MacIntyre D, McConkey P, Khan KM. The effects of proprioceptive or strength training on the neuromuscular function of the ACL reconstructed knee: a randomized clinical trial. Scand J Med Sci Sports. 2003 Apr;13(2):115-23. doi: 10.1034/j.1600-0838.2003.02113.x. PMID 12641643
- [Background] Livesay GA, Rudy TW, Woo SL, Runco TJ, Sakane M, Li G, Fu FH. Evaluation of the effect of joint constraints on the in situ force distribution in the anterior cruciate ligament. J Orthop Res. 1997 Mar;15(2):278-84. doi: 10.1002/jor.1100150218. PMID 9167632
- [Background] Lohmander LS, Ostenberg A, Englund M, Roos H. High prevalence of knee osteoarthritis, pain, and functional limitations in female soccer players twelve years after anterior cruciate ligament injury. Arthritis Rheum. 2004 Oct;50(10):3145-52. doi: 10.1002/art.20589. PMID 15476248
- [Background] Maletius W, Gillquist J. Long-term results of anterior cruciate ligament reconstruction with a Dacron prosthesis. The frequency of osteoarthritis after seven to eleven years. Am J Sports Med. 1997 May-Jun;25(3):288-93. doi: 10.1177/036354659702500303. PMID 9167805
- [Background] Mandelbaum BR, Silvers HJ, Watanabe DS, Knarr JF, Thomas SD, Griffin LY, Kirkendall DT, Garrett W Jr. Effectiveness of a neuromuscular and proprioceptive training program in preventing anterior cruciate ligament injuries in female athletes: 2-year follow-up. Am J Sports Med. 2005 Jul;33(7):1003-10. doi: 10.1177/0363546504272261. Epub 2005 May 11. PMID 15888716
- [Background] Martin-Pintado Zugasti A, Rodriguez-Fernandez AL, Garcia-Muro F, Lopez-Lopez A, Mayoral O, Mesa-Jimenez J, Fernandez-Carnero J. Effects of spray and stretch on postneedling soreness and sensitivity after dry needling of a latent myofascial trigger point. Arch Phys Med Rehabil. 2014 Oct;95(10):1925-1932.e1. doi: 10.1016/j.apmr.2014.05.021. Epub 2014 Jun 10. PMID 24928191
- [Background] Mayoral O, Salvat I, Martin MT, Martin S, Santiago J, Cotarelo J, Rodriguez C. Efficacy of myofascial trigger point dry needling in the prevention of pain after total knee arthroplasty: a randomized, double-blinded, placebo-controlled trial. Evid Based Complement Alternat Med. 2013;2013:694941. doi: 10.1155/2013/694941. Epub 2013 Mar 27. PMID 23606888
- [Background] Myklebust G, Engebretsen L, Braekken IH, Skjolberg A, Olsen OE, Bahr R. Prevention of noncontact anterior cruciate ligament injuries in elite and adolescent female team handball athletes. Instr Course Lect. 2007;56:407-18. PMID 17472324
- [Background] Ordahan B, Kucuksen S, Tuncay I, Salli A, Ugurlu H. The effect of proprioception exercises on functional status in patients with anterior cruciate ligament reconstruction. J Back Musculoskelet Rehabil. 2015;28(3):531-7. doi: 10.3233/BMR-140553. PMID 26406302
- [Background] Postle K, Pak D, Smith TO. Effectiveness of proprioceptive exercises for ankle ligament injury in adults: a systematic literature and meta-analysis. Man Ther. 2012 Aug;17(4):285-91. doi: 10.1016/j.math.2012.02.016. Epub 2012 Mar 27. PMID 22459604
- [Background] Prodromos CC, Han Y, Rogowski J, Joyce B, Shi K. A meta-analysis of the incidence of anterior cruciate ligament tears as a function of gender, sport, and a knee injury-reduction regimen. Arthroscopy. 2007 Dec;23(12):1320-1325.e6. doi: 10.1016/j.arthro.2007.07.003. PMID 18063176
- [Background] Relph N, Herrington L, Tyson S. The effects of ACL injury on knee proprioception: a meta-analysis. Physiotherapy. 2014 Sep;100(3):187-95. doi: 10.1016/j.physio.2013.11.002. Epub 2013 Dec 4. PMID 24690442
- [Background] Saka T. Principles of postoperative anterior cruciate ligament rehabilitation. World J Orthop. 2014 Sep 18;5(4):450-9. doi: 10.5312/wjo.v5.i4.450. eCollection 2014 Sep 18. PMID 25232521
- [Background] Salom-Moreno J, Ayuso-Casado B, Tamaral-Costa B, Sanchez-Mila Z, Fernandez-de-Las-Penas C, Alburquerque-Sendin F. Trigger Point Dry Needling and Proprioceptive Exercises for the Management of Chronic Ankle Instability: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:790209. doi: 10.1155/2015/790209. Epub 2015 Apr 30. PMID 26064172
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Background] Villanueva I, del Mar Guzman M, Javier Toyos F, Ariza-Ariza R, Navarro F. Relative efficiency and validity properties of a visual analogue vs a categorical scaled version of the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index: Spanish versions. Osteoarthritis Cartilage. 2004 Mar;12(3):225-31. doi: 10.1016/j.joca.2003.11.006. PMID 14972339
- [Background] Vrbanic TS, Ravlic-Gulan J, Gulan G, Matovinovic D. Balance index score as a predictive factor for lower sports results or anterior cruciate ligament knee injuries in Croatian female athletes--preliminary study. Coll Antropol. 2007 Mar;31(1):253-8. PMID 17598410
- [Background] Wasmaier J, Kubik-Huch R, Pfirrmann C, Grehn H, Bieg C, Eid K. Proximal anterior cruciate ligament tears: the healing response technique versus conservative treatment. J Knee Surg. 2013 Aug;26(4):263-71. doi: 10.1055/s-0032-1329720. Epub 2012 Dec 20. PMID 23258320
- [Background] Bron C, de Gast A, Dommerholt J, Stegenga B, Wensing M, Oostendorp RA. Treatment of myofascial trigger points in patients with chronic shoulder pain: a randomized, controlled trial. BMC Med. 2011 Jan 24;9:8. doi: 10.1186/1741-7015-9-8. PMID 21261971
- [Background] Pecos-Martin D, Montanez-Aguilera FJ, Gallego-Izquierdo T, Urraca-Gesto A, Gomez-Conesa A, Romero-Franco N, Plaza-Manzano G. Effectiveness of dry needling on the lower trapezius in patients with mechanical neck pain: a randomized controlled trial. Arch Phys Med Rehabil. 2015 May;96(5):775-81. doi: 10.1016/j.apmr.2014.12.016. Epub 2015 Jan 9. PMID 25582412
- [Background] Mason JS, Tansey KA, Westrick RB. Treatment of subacute posterior knee pain in an adolescent ballet dancer utilizing trigger point dry needling: a case report. Int J Sports Phys Ther. 2014 Feb;9(1):116-24. PMID 24567862